CLINICAL TRIAL: NCT06333262
Title: A Phase 2 Study of Fixed Duration Therapy With Pirtobrutinib and Obinutuzumab in Previously Untreated Chronic Lymphocytic Leukemia (POP)
Brief Title: Fixed Duration Pirtobrutinib and Obinutuzumab in Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inhye Ahn (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Inhye Ahn, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-017
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Bruton's tyrosine kinase inhibitor; Pirtobrutinib; Obinutuzumab; Fixed-duration
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib-Obinutuzumab (Experimental): Eligible participants will receive initial treatment with pirtobrutinib and obinutuzumab for 12 cycles. Participants with progressive chronic lymphocytuc leukemia or small lymphocytic lymphoma during the off-treatment follow-up will receive continuous pirtobrutinib monotherapy.
  Interventions: Drug: Pirtobrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Pirtobrutinib — Initial treatment:
  - Pirtobrutinib 200 mg by mouth (PO) daily from Cycle 1 Day 1 until the end of Cycle 12. Each cycle is 28 days.
  Re-treatment:
  -Pirtobrutinib 200 mg PO daily continuously
Drug: Obinutuzumab — Obinutuzumab is given intravenously from Cycle 7 to Cycle 12, for total 6 cycles during initial treatment only.
  Initial treatment:
  - Obinutuzumab intravenous (IV) following the standard schedule from Cycle 6 through Cycle 12 (total 6 cycles: 100 mg on Cycle 6 Day 1, 900 mg on Cycle 6 Day 2, 1000 mg on Cycle 6 Day 8 and Cycle 6 Day 15, 1000 mg on Day 1 of Cycle 7 through Cycle 12).

SUMMARY:
This study will evaluate fixed-duration therapy with pirtobrutinib and obinutuzumab given over 12 cycles (approximately 1 year) as first-line treatment of chronic lymphocytic leukemia or small lymphocytic lymphoma (CLL or SLL).

DETAILED DESCRIPTION:
This is an open-label, multicenter, single-arm phase 2 study of pirtobrutinib with obinutuzumab for participants with CLL or SLL. Eligible participants will receive 6 cycles of pirtobrutinib alone followed by an additional 6 cycles of pirtobrutinib-obinutuzumab combination therapy. All participants will stop treatment after 12 cycles in total (approximately 1 year).

If CLL progresses and requires treatment after 1-year of therapy, participants will receive retreatment with pirtobrutinib only. Participants will be followed for up to a total of 10 years. Up to 60 participants will take part in this study.

The U.S. Food and Drug Administration (FDA) has approved pirtobrutinib for continuous treatment of CLL that has relapsed or become refractory to other treatments. Pirtobrutinib is not approved for the first-line treatment of CLL/SLL nor for fixed-duration therapy. The FDA has approved obinutuzumab for the treatment of CLL.

The research study procedures include screening for eligibility, study treatment visits, electrocardiograms, imaging (e.g. computerized tomography or CT scans), blood tests, saliva tests, bone marrow biopsies, and/or lymph node biopsies (if feasible).

Loxo Oncology at Eli Lilly and Company is supporting this study by providing pirtobrutinib and research funding.

ELIGIBILITY:
Key Inclusion Criteria:

* Meet 2018 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines for the diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL).
* Presence of measurable disease (absolute lymphocyte count > 5,000/µL, palpable or measurable lymph nodes ≥1.5cm on imaging, or bone marrow involvement of CLL ≥ 30%).
* No prior systemic therapy for CLL or SLL.
* Currently have an indication for treatment as defined by the following 2018 IWCLL guidelines
* Age ≥ 18 years
* Eastern Cooperative Oncology Group performance status ≤ 2
* Adequate organ and bone marrow function as defined by the study protocol
* Ability to take oral medications.
* Ability to understand and the willingness to sign a written informed consent document.

Key Exclusion Criteria:

* Known or suspected Richter's transformation or known central nervous system involvement.
* History of bleeding disorders
* History of stroke or intracranial hemorrhage within 6 months of starting study therapy.
* Significant cardiovascular disease such as uncontrolled arrhythmia, Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction < 40% by any methods in the 12 months prior to study therapy.
* History of other malignancies with life expectancy of < 2 years.
* Receiving any other investigational agents.
* Concurrent systemic immunosuppression < 28 days of study therapy or administration of > 20 mg of prednisone or equivalent daily < 7 days of study therapy.
* Vaccinated with live vaccine within 4 weeks of starting study therapy.
* Major surgery within 4 weeks of starting study therapy.
* Ongoing or recent infection requiring intravenous antimicrobials at time of screening. Prophylactic antibiotics are allowed if there is no evidence of active infection and the antibiotics is not included on the list of the prohibited medications.
* Patients who have tested positive for HIV are excluded due to potential drug-drug interactions between anti-retroviral medications and pirtobrutinib and risk of opportunistic infections with both HIV and irreversible BTK inhibitors. For patients with unknown HIV status, HIV testing will be performed at Screening and result should be negative for enrollment.
* Active human T cell leukemia virus infection or active hepatitis B or C virus infection
* Known active cytomegalovirus infection
* Pregnancy, lactation or plan to breastfeed during the study or within 6 months of the last dose of study treatment.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug
* Active uncontrolled auto-immune cytopenia.
* Significant co-morbid condition or disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response after initial therapy | 1 year since treatment initiation
  Defined by the 2018 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines

SECONDARY OUTCOMES:
Overall response rate | 1 year since treatment initiation
  Defined by the 2018 IWCLL guidelines
Rate of partial response | 1 year since treatment initiation
  Defined by the 2018 IWCLL guidelines
Time to next line of therapy | 5 years after the last enrollment
  Time from the initiation of study therapy until the next line of therapy (excluding pirtobrutinib re-treatment)
Event-free survival | 5 years after the last enrollment
  Time from the initiation of study therapy until pre-defined events (progression, death, or start of a new treatment)
Progression-free survival | 5 years after the last enrollment
  Time from the initiation of study therapy until disease progression or death
Overall survival | 5 years after the last enrollment
  Time from the initiation of study therapy until death
Rate of re-treatment with pirtobrutinib | 5 years after the last enrollment
  Rate of re-treatment with pirtobrutinib on study

CONTACTS AND LOCATIONS:
Overall Officials: Inhye E Ahn, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - New England Cancer Specialists, Scarborough, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu